CLINICAL TRIAL: NCT04855565
Title: Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Subcutaneous Doses of ALY688-SR in Generally Healthy Overweight or Obese Adults
Brief Title: ALY688-SR in Generally Healthy Overweight or Obese Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inability to recruit due to COVID-19 pandemic restrictions
Sponsor: Allysta Pharmaceutical (Industry)
Collaborators: INC Research Australia Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALY688-SR-101
Record Dates: First submitted 2021-04-16; First posted 2021-04-22 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Single dose escalation study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Site staff treating subjects, subjects themselves and the Investigator will be blinded to the treatments being administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALY688-SR (Active Comparator): single dose subcutaneous injection
  Interventions: Drug: ALY688-SR
- Matching placebo for ALY688-SR (Placebo Comparator): single dose subcutaneous injection
  Interventions: Drug: ALY688-SR

INTERVENTIONS:
Drug: ALY688-SR — single dose subcutaneous injection

SUMMARY:
First in human study of ALY688-SR administered as a subcutaneous injection

DETAILED DESCRIPTION:
The study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single ascending doses of ALY688-SR compared to placebo administered as a subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 24 to 35 kg/m2 Body weight 60 to 120 kg,

Exclusion Criteria:

* Confirmed diabetes on treatment Inadequately managed hypertension Poorly controlled hypercholesterolemia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Change between pre- and post-intervention safety and tolerability assessments | baseline, pre-intervention through study completion at 16 days
  Incidence of Treatment-Emergent Adverse Events as assessed by lab evaluations, ECG, vital signs and physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Ben Snyder, MD, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No